CLINICAL TRIAL: NCT05906823
Title: Metabonomics for Distinguishing Between Benign and Malignant Pleural Effusion and Assessing the Prognosis of Lung Cancer Patients With Malignant Pleural Effusion
Brief Title: Analysis of Metabonomics for Pleural Effusion
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XHJY20230508
Record Dates: First submitted 2023-05-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Pleural Diseases
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — pleural effusion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- benign pleural effusion: Patients with benign pleural effusion.
  Interventions: Other: Detection of pleural effusion
- malignant pleural effusion patients with bad prognosis: The OS time of malignant pleural effusion patients is<1 year.
  Interventions: Other: Detection of pleural effusion
- malignant pleural effusion patients with good prognosis: The OS time of malignant pleural effusion patients is ≥1 year.
  Interventions: Other: Detection of pleural effusion

INTERVENTIONS:
Other: Detection of pleural effusion — Detection of pleural effusion

SUMMARY:
This is a multicenter retrospective study that collected diagnostic information of patients with pleural effusion. The overall survival (OS) time of malignant patients was followed up, defined as the time from diagnosis to death. Clinical data and residual pleural effusion specimens were collected from patients. Metabonomics was utilized to differentiate between benign and malignant pleural effusion and to evaluate the prognosis of lung cancer patients with malignant pleural effusion.

DETAILED DESCRIPTION:
Pleural effusion (PE) is a common yet challenging problem in clinical settings. PE is a symptom caused by over 50 diseases and is typically classified as either malignant pleural effusion (MPE) or benign pleural effusion (BPE). MPE affects a significant number of individuals, with an estimated annual incidence of 500-700 cases per million population. Metastatic cancer is the leading cause of MPE, and lung cancer accounts for approximately 37.5% of cases. The management of MPE is a major clinical challenge due to its association with a typically poor prognosis, with a median survival of only 3 to 12 months. However, predicting survival in MPE patients can be difficult due to significant heterogeneity in underlying malignancy and patient performance status. Therefore, accurate prognostication remains a significant challenge in the management of MPE.

Metabonomics is an analytical technique for detecting metabolites in biological samples and has been widely used in disease diagnosis and prognosis evaluation in recent years. The aim of this study is to use Metabonomics technology to compare and analyze the differences in metabolites between benign and malignant pleural effusion, and to explore its application in the prognosis evaluation of lung cancer patients with malignant pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 80 Years; detection of pleural effusion by chest computed tomography, radiography, or ultrasonography; pathologically confirmed lung cancer in pleural effusion.

Exclusion Criteria:

* pleural effusion not caused by lung cancer or of unknown origin; other concurrent malignant diseases; incomplete information; lack of any follow-up data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pleural effusion
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Metabolomic detection of pleural effusion to distinguish between benign and malignant pleural effusion | Within two weeks of detection of a pleural effusion
  The concentration of metabolites in the sample of pleural effusion of benign and malignant pleural effusion patients.

SECONDARY OUTCOMES:
Predicting one-year survival prognosis in patients with malignant pleural effusion | 1 year
  Number of Patients with malignant pleural effusion followed up for 1 year after diagnosis to collect survival information.

IPD SHARING:
Plan to Share IPD: No